CLINICAL TRIAL: NCT06705049
Title: Retrospective Study on Leptomeningeal Metastasis of Solid Tumors
Status: Enrolling by invitation | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2024687
Record Dates: First submitted 2024-11-21; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Leptomeningeal Metastasis
MeSH Terms: conditions — Meningeal Carcinomatosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: MRI — On MRI, some lesions present as linear enhancement, while others exhibit nodular enhancement

SUMMARY:
The goal of this observational study is to investigate the clinical characteristics, treatment outcomes, and prognostic factors of leptomeningeal metastasis (LM), a serious complication of advanced cancer. LM occurs when tumor cells spread to the leptomeninges and subarachnoid space, leading to neurological symptoms and poor prognosis. This study aims to answer:

What are the common clinical features of LM? How do different treatments affect survival and quality of life? What factors influence patient outcomes?

Background With advancements in cancer treatment, patient survival has improved significantly, but late-stage complications like LM are becoming more common. LM is seen in about 5% of patients with metastatic cancers such as lung cancer, breast cancer, and melanoma. Symptoms can range from mild headaches and nausea to severe neurological issues, including vision loss, hearing impairment, or limb weakness, making LM challenging to diagnose and treat.

Diagnosis often involves MRI with gadolinium enhancement and cerebrospinal fluid (CSF) analysis. Treatment options include intrathecal chemotherapy, targeted therapy, radiotherapy, and supportive care. However, LM remains a condition with poor prognosis, and there are no standardized treatment guidelines.

Study Design This study will retrospectively review LM cases treated at our hospital. Data will include: Patient demographics (age, gender, cancer type)Symptoms and clinical findings Treatment types (e.g., chemotherapy, targeted therapy, radiotherapy) Survival outcomes and factors influencing prognosis

Hypothesis The findings from this study aim to provide better insight into LM's clinical characteristics and treatment outcomes. This will help guide more effective, individualized treatment approaches and improve quality of life for patients with LM.

DETAILED DESCRIPTION:
Experimental Procedure：

1. Case Collection This study collected all cases of leptomeningeal metastasis (LM) diagnosed through cerebrospinal fluid cytology at our center between January 2014 and August 2024. The collected data includes:Demographic information: Age, gender Clinical presentation: Chief complaints, current medical history, past medical history Pathological data: Pathology reports Laboratory findings: Blood lipids, renal function, platelet counts Physical characteristics: Body mass index (BMI), smoking history Surgical records: Detailed records of any surgeries Imaging data: Preoperative, postoperative, and follow-up imaging studies Survival data: Patient survival status and outcomes
2. Data Collection Methods Follow-up and Survival Information

   Survival data and follow-up information were collected via telephone interviews with patients or their families.

   Medical History and General Information

   Current medical history, past medical history, and other general information were extracted from hospital inpatient medical records.

   Imaging Data

   Imaging data, including preoperative, postoperative, and follow-up imaging studies, were retrieved and copied from the hospital's Picture Archiving and Communication System (PACS).
3. Statistical Analysis

   All collected data were subjected to statistical analysis to evaluate trends, correlations, and factors influencing patient outcomes. Specific statistical methods include:

   Descriptive statistics to summarize demographic and clinical characteristics Inferential statistics to analyze potential associations between variables and survival outcomes Multivariate regression models to identify prognostic factors
4. Study Design and Ethical Considerations This study is a retrospective, observational study. It does not involve any intervention or sample collection from patients. All data were collected from existing medical records, imaging systems, and follow-up interviews, ensuring no additional burden on patients.

By adhering to these methods, the study aims to provide insights into the clinical characteristics and survival outcomes of LM patients while maintaining ethical and methodological rigor.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a previously or recently diagnosed solid tumor in other parts of the body.
2. Detection of metastatic tumor cells in cerebrospinal fluid (CSF) cytology examination.
3. The patient has signed an informed consent form for the donation of biological samples and health-related information.
4. Age between 18 and 80 years.
5. The participant is willing to take part in this study.

Exclusion Criteria:

1. Presence of a clearly defined single intracranial lesion with a mass effect.
2. Pregnancy or breastfeeding.
3. Any other conditions deemed unsuitable for participation in this clinical trial, as evaluated by the physician.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with leptomeningeal metastases
Sampling Method: Non-Probability Sample
Enrollment: 107 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 2024/01/01-2024/08/31
  The survival period from the time of diagnosis of leptomeningeal metastases (LM) to the time of death.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Xie, Study Director — Fudan University
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
no relative sharing plan